CLINICAL TRIAL: NCT01856556
Title: A Randomized, Double-Blind, Placebo-Controlled Single Intravenous and Oral Ascending Dose Study of the Safety, Tolerability and Pharmacokinetics of NRX-1074 in Normal Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of NRX-1074 in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRX1074-C-101
Record Dates: First submitted 2013-05-13; First posted 2013-05-17 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: safety; tolerability; pharmacokinetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- NRX-1074, 1 mg (Experimental): 1 mg IV
  Interventions: Drug: NRX-1074
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo
- NRX-1074, 5 mg (Experimental): 5 mg IV
  Interventions: Drug: NRX-1074
- NRX-1074, 10 mg IV (Experimental): 10 mg
  Interventions: Drug: NRX-1074
- NRX-1074, 50 mg IV (Experimental): 50 mg
  Interventions: Drug: NRX-1074
- NRX-1074, 25 mg PO (Experimental): 25 mg
  Interventions: Drug: NRX-1074
- NRX-1074, 125 mg PO (Experimental): 125 mg
  Interventions: Drug: NRX-1074

INTERVENTIONS:
Drug: NRX-1074 — Single IV or PO administration
  Other Names: NMDA receptor functional glycine-site partial agonist
  Arms: NRX-1074, 1 mg; NRX-1074, 10 mg IV; NRX-1074, 125 mg PO; NRX-1074, 25 mg PO; NRX-1074, 5 mg; NRX-1074, 50 mg IV
Drug: Placebo — Single IV or PO placebo administration
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of a single intravenous (IV) and oral (PO) ascending dose of NRX-1074 as evidenced by the incidence and severity of adverse events (AEs), changes in serum chemistry, hematology, and urinalysis, changes in physical examination findings and subject-reported symptoms.

The secondary objectives of this study are to assess the plasma and cerebrospinal fluid (CSF) pharmacokinetics (PK), the oral bioavailability of experimental formulations and the renal elimination through urine concentration of NRX-1074 through 24 hours following dosing.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, single ascending dose level study. On Day 1, eligibility of each subject will be confirmed, physical examination will be performed, and blood and urine for laboratories will be obtained. Each subject will be randomized, then will receive either a single IV, SC or IN dose of GLYX-13 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects
2. Aged 18 to 55 years
3. For female subjects, surgically sterile or at least 2 years menopausal, or using an acceptable method of birth control from date of screening to at least 30 days after the last dose of study drugIf of childbearing potential, have a documented negative blood or urine pregnancy test within 24 hours prior to dosing.
4. Clinical laboratory values less than or equal to 2 times the upper limit of normal (ULN) or deemed not clinically significant by the Investigator.
5. Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Observed and laboratory-confirmed safety | 28 days

SECONDARY OUTCOMES:
Plasma concentration of parent drug will be assessed over time to estimate duration of pharmacodynamics in future efficacy trials. Plasma concentration and pharmacokinetics will be related in time to observed side effects. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Grace Ting, MD, Principal Investigator — Lotus Clinical Research
Locations (1):
- Lotus Clinical Research, Pasadena, California, United States